CLINICAL TRIAL: NCT05386602
Title: Development and Validation of a Patient Reported Experience Measure for Experimental Cancer Medicine (PREM-ECM)
Brief Title: Development and Validation of a Patient Reported Experience Measure for Experimental Cancer Medicine
Acronym: PREM-ECM
Status: Completed | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18_CPCR_15
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2023-08

CONDITIONS: Cancer
Keywords: Patient Experience; Experimental Medicine; Patient Reported Experience Measure; PREM
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Prior trial patients: In stage III, patients who have been on an experimental cancer medicine trial for less than six weeks will complete a draft PREM-ECM (less than six weeks), the EORTC PATSATC33 and HAD questionnaires at entry to the PREM study (baseline/time point 1 (T1)). Approximately 50 patients will be asked to repeat the draft of the PREM-ECM (less than six weeks) approximately one week later at time point 2 (T2). In stage IV, the PREM-ECM will be administered alone.
- On trial patients: In stage III, patients who have been on an experimental cancer medicine trial for more than six weeks will complete a draft PREM-ECM (more than six weeks), the EORTC PATSATC33 and HAD questionnaires at entry to the PREM study (baseline/time point 1 (T1)). Approximately 50 patients will be asked to repeat the draft of the PREM-ECM (more than six weeks) approximately one week later at time point 2 (T2). In stage IV, the PREM-ECM will be administered alone.
- Carers of patients: In stage III, carers of patients recruited on an experimental cancer medicine trial will be asked to complete a draft PREM-ECM-carers, the Adult Carer Quality of Life Questionnaire (AC-QOL), the EQ5D-5L, and the Hospital Anxiety and Depression Scale (HADS) at entry to the PREM study (baseline/time point 1 (T1)). Approximately 50 carers will be asked to repeat the draft of the PREM-ECM-carers approximately one week later at time point 2 (T2). In Stage IV, the PREM-ECM-carer will be administered alone.

SUMMARY:
This is a four stage, non-interventional study to develop and pilot test a Patient Reported Experience Measure (PREM) in experimental cancer medicine trials.

DETAILED DESCRIPTION:
PREM-ECM will be conducted in four stages

Stage I - Item generation Two focus groups with four-eight participants each and approximately 20 interviews will be conducted with experimental cancer medicine trial participants to capture their experiences of participating in clinical trials and the care they have received during screening and trial participation. The investigators will also conduct up to ten interviews with informal carers (either as dual carer-patient or carer only interviews). Potential items for PREM-ECM inclusion will be extracted from these interviews (depending on carer data extraction their views will be incorporated into the patient item list or a separate 'carer experience' item list. Participants in Stage I will be asked to consent to possible cognitive interviews later in stage II. Interviews will be audio recorded using a Dictaphone which encrypts files in real time.

Stage II - Cognitive interviewing Following the creation of a draft item list, approximately five-seven participants from Stage I and three-five study naïve patients will undergo cognitive interviews to ensure that all items are clear and easily understood. Interviews will be audio recorded using a Dictaphone which encrypts files in real time.

Stage III - Item reduction and refinement for two PREM-ECMs A draft PREM-ECM (less than six weeks) and the EORTC PATSATC33 and HAD questionnaires will be administered to approximately 180 participants recruited into an experimental cancer medicine trial at entry to the PREM study (baseline/time point 1 (T1)). Approximately 50 patients will be asked to repeat the draft of the PREM-ECM (less than six weeks) approximately one week later at time point 2 (T2) - this is to test for individual item test retest reliability. A draft of the PREM-ECM (over six weeks) and the EORTC PATSATC33 and HAD questionnaires will be administered to approximately 180 participants recruited into an experimental cancer medicine trial at entry to the PREM study (baseline/time point 1 (T1)). Approximately 50 patients will be asked to repeat the PREM-ECM during approximately one week later at time point 2 (T2) - this is to test for individual item test retest reliability.

A draft PREM-ECM-carers, the Adult Carer Quality of Life Questionnaire (AC-QOL), the EQ5D-5L, and the Hospital Anxiety and Depression Scale (HADS) questionnaire will be administered to approximately 150 carers of patients recruited into an experimental cancer medicine trial (baseline/time point 1 (T1)). Approximately 50 carers will be asked to repeat the draft of the PREM-ECM - carers approximately one week later at time point 2 (T2) - this is to test for retest reliability.

Stage IV - Pilot testing of the PREM-ECM Both the PREM-ECM will be pilot tested with approximately 20 patients per questionnaire at The Christie site to assess its feasibility for routine collection of patient experience data.

ELIGIBILITY:
Patient Inclusion Criteria:

* Recruited into a phase 1-2 experimental cancer medicine clinical trial
* Ability to understand and communicate in the English language
* Able to provide written informed consent

Patient Exclusion Criteria:

* Patients who are not able to complete informed consent or the study questionnaires

Carer Inclusion Criteria:

* Ability to understand and communicate in the English language
* Able to provide written informed consent
* Nominated by the patient as their primary caregiver/most able to describe relevant experience

Carer Exclusion Criteria:

* Carers who are not able to complete informed consent or the study questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients and carers of patients who are recruited into a phase 1-2 experimental cancer medicine clinical trial. Patients and carers will be identified by their treating clinician/physician or another healthcare professional at the hospital recruitment site.
Sampling Method: Non-Probability Sample
Enrollment: 570 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Patients reported care experience | 1 week
  Collected by a Patient Reported Experience Measure in Experimental Cancer Medicine (PREM-ECM) questionnaire. A five point Likert scale is used to specify their levels of agreement with a statement, from low (1) to high (5). Higher scores are interpreted as better patient experience.
Patient quality of life | 1 week
  European Organisation Research and Treatment of Cancer (EORTC) Satisfaction with cancer care core questionnaire (PATSATC33). incorporates seven multi-item scales to assess doctors' technical skills, information exchange and affective behaviour, nurses/radiotherapy technicians' information/responsiveness and affective behaviour, and services and care organisation in terms of coordination and interaction with health care providers. In addition, five single items assess family/close persons' care involvement, access, environment, and overall perceived care quality. All of the scales and single-item measures range in score from 0 to 100. A high score represents a high level of satisfaction with care / perceived care quality.
Patient anxiety and depression | 1 week
  Hospital Anxiety and Depression Scale (HADS). It comprises 14 items, seven to assess anxiety (HADS-A), namely items 1, 3, 5, 7, 9, 11, and 13; and seven to assess depression (HADS-D), namely items 2, 4, 6, 8, 10, 12, and 14. Each item receives a score from 0 to 3 on a Likert Scale. The total score for each HADS-A and HADS-D scale is obtained by adding the individual scores for each item, with the maximum score 21. The presence or absence of depression and anxiety was defined, for each respective scale, based on the following cutoff values: HADS (anxiety): 0-8 equal to (=) no anxiety; greater than (>) 9 = anxiety; HADS (depression): 0-8 = no depression; >9 = depression.
Carer quality of life | 1 week
  Adult Carer Quality of Life Questionnaire (AC-QOL). It is made up of eight different areas (care giving, caring preference, patient care stress, financial issues, personal development, valuing, caregiving ability and caregiver satisfaction). In scale evaluation, 0-40 points indicate "low quality of life", 41-80 points "average quality of life" and 81-120 points indicate "high quality of life"
Carer health-related quality of life | 1 week
  EQ-5D-5L. Consists of two components: a health state profile and a visual analog scale (VAS). EQ-5D health state profile comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. The 5D-5L systems are converted into a single index utility score between 0 to 1, where a higher score indicates a better health state. The VAS records the participant's health on a 0-100 mm VAS scale, with 0 indicating "the worst health you can imagine" and 100 indicating "the best health you can imagine". Higher scores of EQ VAS indicate better health.
Carer reported care experience | 1 week
  Collected by a Patient Reported Experience Measure in Experimental Cancer Medicine- Carers (PREM-Carers) questionnaire. A five point Likert scale is used to specify their levels of agreement with a statement, from low (1) to high (5). Higher scores are interpreted as better carer experience.
Carer anxiety and depression | 1 week
  Hospital Anxiety and Depression Scale (HADS). It comprises 14 items, seven to assess anxiety (HADS-A), namely items 1, 3, 5, 7, 9, 11, and 13; and seven to assess depression (HADS-D), namely items 2, 4, 6, 8, 10, 12, and 14. Each item receives a score from 0 to 3 on a Likert Scale. The total score for each HADS-A and HADS-D scale is obtained by adding the individual scores for each item, with the maximum score 21. The presence or absence of depression and anxiety was defined, for each respective scale, based on the following cutoff values: HADS (anxiety): 0-8 equal to (=) no anxiety; greater than (>) 9 = anxiety; HADS (depression): 0-8 = no depression; >9 = depression.

CONTACTS AND LOCATIONS:
Overall Officials: Sally Taylor, PhD, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results/Publication — https://doi.org/10.1186/s12885-024-11963-x